CLINICAL TRIAL: NCT01637753
Title: Phase 3 Study of Carmustine Sustained Release Implant (CASANT) to Treat Recurrent Malignant Glioma
Brief Title: Safety and Efficacy Study of Intracranially Implanted Carmustine to Treat Recurrent Malignant Glioma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Lanjin Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LJ-Glioma 3.1.0 Version
Record Dates: First submitted 2012-07-04; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Oligoastrocytoma; Glioblastoma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma | interventions — Carmustine; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carmustine Sustained Release Implant (Experimental)
  Interventions: Drug: Carmustine(BCNU)
- Surgical control group (Sham Comparator)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: Carmustine(BCNU) — Carmustine Sustained Release Implant
  Other Names: BCNU
  Arms: Carmustine Sustained Release Implant
Procedure: Surgery — Routine tumor resection surgery
  Arms: Surgical control group

SUMMARY:
The purpose of the study is to determine the safety and efficacy of intracranially implanted Carmustine in the treatment of patients with recurrent malignant glioma.

DETAILED DESCRIPTION:
Malignant gliomas recur mostly 2 cm within originated area. Local therapies therefore become particular important. Gliadel wafer developed in the States and marketed in the developed countries is an example of such treatments. The product in this study, Carmustine Sustained Release Implant (CASANT), is similar to that of Gliadel wafer as for the API(Active Pharmaceutical Ingredient), but different as for drug delivering system. As required, the preliminary clinical studies were conducted in China. Based on the results of phase I/II , 8-10 wafers containing given dose of BCNU will be administered intracranially in this phase III to the tumor resected cavity to investigate the safety and efficacy in the treatment of recurrent malignant glioma in 212 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 to 70 years old, signed ICF;
* At least 4 weeks after previous chemotherapy (6 weeks since nitrosoureas);
* KPS ≥ 60;
* Unilateral, Supratentorial, solitary lesion and not crossing the midline(exclude patients with little tumors near the resectable tumor even if investigators think they are single lesions)
* No obvious important organ dysfunction: Blood routine: White blood cell (WBC) ≥ 4.0×109/L, Absolute neutrophil count (ANC)≥ 1.5×109/L, Platelets≥ 100×109/L, Hemoglobin≥ 90 g/L; Hepatic function:Serum total bilirubin ≤1.5 times upper limit of laboratory normal; Aspartate aminotransferase (AST) and/or Alanine aminotransferase (ALT)<2.5 times upper limit of laboratory normal; Renal function:Serum creatinine ≤1.5 times upper limit of laboratory normal;
* Not Pregnant or lactating for women of childbearing potential.

Exclusion Criteria:

* Tumor located at ventricular system, Open ventricle tumor cavity postoperatively;
* Concomitant with other life-threatening diseases and with life expectancy <3 months;
* Allergic to nitrosourea drugs;
* With history of intracranial radiotherapy or implant chemotherapy;
* With serious cardiac, pulmonary, hepatic and renal dysfunction, poor glycemic control;
* Investigators thought unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 12 months

SECONDARY OUTCOMES:
Overall Survival Rate | 12 months
Progress Free Survival Rate at 6 months | 12 months
Tumor response rate | 12 months
KPS Score | 12 months
QOL Score | 12 months
Safety of intracranially implanted carmustine after maximal tumor resection | 12 months
  Occurrence rate of adverse event and serious adverse event revealed by laboratory test outcomes including blood routine and chemistry as well as physical examination, vital signs including blood presure, temperature, respiratory rate , heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong P Chen, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangzhou, China